CLINICAL TRIAL: NCT02545023
Title: Supportive Care Needs of Breast Cancer Survivors: A Needs Assessment
Brief Title: Supportive Care Questionnaires in Gathering Data on Unmet Needs and Health-Related Quality of Life in Latina Breast Cancer Survivors After Surgery, Chemotherapy, or Radiation Therapy
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1B-15-3; NCI-2015-01389 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-15-00487; 1B-15-3 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-09-06; First posted 2015-09-09 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Breast Carcinoma; Cancer Survivor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (Supportive care, health-related QOL): Participants complete the demographic questionnaire, SCNS-34, SF-36, and the Lifestyle Needs Survey. Within 1 year of completing questionnaires, some participants may complete a one-hour in-person one-on-one interview comprising questions about the challenges and experiences of cancer survivorship, their health and well-being, and supportive care needs.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Complete an in-person one-on-one interview
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete the demographics questionnaire, SCNS-34, SF-36, and Lifestyle Needs Survey

SUMMARY:
This phase I/II research trial studies supportive care questionnaires in gathering data on unmet needs and health-related quality of life in Latina breast cancer survivors after surgery, chemotherapy, or radiation therapy. Questionnaires that address unmet supportive care needs and health-related quality of life of breast cancer survivors may help doctors learn about barriers to cancer care that are linked to language, acculturation, knowledge about diagnosis and care, and financial concerns. Learning about unmet needs of breast cancer patients may help increase quality of life and decrease healthcare utilization and costs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the supportive care needs and preferences of breast cancer survivors at Los Angeles County + University of Southern California (USC) Medical Center (LAC+USC).

SECONDARY OBJECTIVES:

I. To determine the lifestyle-related challenges of individuals with breast cancer being treated at LAC+USC.

II. To determine the communication and healthcare delivery style needs and preferences of individuals with breast cancer being treated at LAC+USC.

OUTLINE:

Participants complete the demographic questionnaire, Supportive Care Needs Survey (SCNS)-34, 36-item Short Form Health Survey (SF-36), and the Lifestyle Needs Survey. Within 1 year of completing questionnaires, some participants may complete a one-hour in-person one-on-one interview comprising questions about the challenges and experiences of cancer survivorship, their health and well-being, and supportive care needs.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving ongoing care, including routine follow-up, at LAC+USC
* Diagnosis of breast cancer
* Completed primary surgical treatment, chemotherapy, and/or radiation
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Inability to sign written informed consent or to complete questionnaires/surveys
* Diagnosis of metastatic cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Latina breast cancer survivors receiving ongoing care, including routine follow-up, at LAC+USC.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Lifestyle-related supportive care needs and preferences in breast cancer patients at LAC+USC, as measured by the Lifestyle Needs Survey and interview | Up to 1 year
  For descriptive purposes, means, standard deviations, frequencies, and percentages will be calculated for each survey measure as well as for demographic variables. The remaining statistical analysis will consist of a comparison of HRQOL and all SNCS-34 domains. Correlation coefficients between SF-36 total score and total score of each SNCS domain will be calculated. All analyses will be conducted using a two-tailed test at the 0.05 significance level.
Supportive care needs and preferences of breast cancer survivors at LAC+USC, as measured by the SCNS-34, Lifestyle Needs Survey, and interview | Up to 1 year
  For descriptive purposes, means, standard deviations, frequencies, and percentages will be calculated for each survey measure as well as for demographic variables. The remaining statistical analysis will consist of a comparison of HRQOL and all SNCS-34 domains. Correlation coefficients between SF-36 total score and total score of each SNCS domain will be calculated. All analyses will be conducted using a two-tailed test at the 0.05 significance level.

SECONDARY OUTCOMES:
Communication and healthcare delivery style needs and preferences of individuals with breast cancer being treated at LAC+USC, as measured by the Lifestyle Needs Survey | Up to 1 year
  For descriptive purposes, means, standard deviations, frequencies, and percentages will be calculated for each survey measure as well as for demographic variables. The remaining statistical analysis will consist of a comparison of HRQOL and all SNCS-34 domains. Correlation coefficients between SF-36 total score and total score of each SNCS domain will be calculated. All analyses will be conducted using a two-tailed test at the 0.05 significance level.
Lifestyle-related challenges of individuals with breast cancer being treated at LAC+USC, as measured by the Lifestyle Needs Survey and interview | Up to 1 year
  For descriptive purposes, means, standard deviations, frequencies, and percentages will be calculated for each survey measure as well as for demographic variables. The remaining statistical analysis will consist of a comparison of HRQOL and all SNCS-34 domains. Correlation coefficients between SF-36 total score and total score of each SNCS domain will be calculated. All analyses will be conducted using a two-tailed test at the 0.05 significance level.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Sleight, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States